CLINICAL TRIAL: NCT00123552
Title: Longitudinal Comparison of Combination Antimalarial Therapies in Ugandan Children: Evaluation of Safety, Tolerability, and Efficacy
Brief Title: Longitudinal Antimalarial Combinations in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Rosenthal, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-068; UCSF-CHR Number:H2397-25789-01
Record Dates: First submitted 2005-07-22; First posted 2005-07-25 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Malaria
Keywords: Uganda, malaria, combination antimalarial therapy
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Pyrimethamine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Amodiaquine+Artesunate
- 2 (Experimental)
  Interventions: Drug: Amodiaquine+Sulfadoxine/Pyrimethamine
- 3 (Experimental)
  Interventions: Drug: Artemether+Lumefantrine

INTERVENTIONS:
Drug: Amodiaquine+Artesunate — Amodiaquine 10 mg/kg on day 1, then 5 mg/kg on day 2 and 3; Artesunate 4 mg/kg/d for three days
  Arms: 1
Drug: Amodiaquine+Sulfadoxine/Pyrimethamine — Amodiaquine 10 mg/kg on day 1, then 5 mg/kg on day 2 and 3; S/P at 25 mg/kg sulfadoxine and 1.25 mg/kg pyrimethamine single dose
  Arms: 2
Drug: Artemether+Lumefantrine — Artemether 20 mg + Lumefantrine 120 mg 6 dose regimen at 0 and 8 hours on day 1 and twice daily on days 2 and 3:5 kg to < 15 kg: 1 tab/dose; 15 to 24 kg: 2 tabs/dose; >35 kg:4 tabs per dose
  Arms: 3

SUMMARY:
The purpose of this study is to compare different ways of treating uncomplicated malaria in a group of Ugandan children. The study will be divided into 2 parts. Part 1 of the study will consist of 600 children, ages 1-10, living in the Mulago III Parish of Kampala. Approximately 90 children living in the same household as children from the Phase 1 portion of the study will be enrolled in Phase II of this study. Participants in Phase II of the study will receive an insecticide treated net to cover their bed. Over the course of the study, participants will be tested for malaria when they present to the clinic with a fever or illness. Participants that test positive for malaria will be given 1 of 3 possible study drug combinations. Study procedures will include physical exams and blood samples. Children will participate for about 3 years. Protocol 05-0110 is a study related to this protocol.

DETAILED DESCRIPTION:
Malaria is one of the most important infectious diseases worldwide. New therapies are needed, and it is generally agreed that combination therapy for uncomplicated malaria offers the best opportunity for effective therapy and for the prevention of selection of resistant parasites. Phase I of this study will be a randomized, single-blinded longitudinal clinical trial, comparing the efficacies of different combination antimalarial regimens for the treatment of uncomplicated malaria in a cohort of Ugandan children. The clinical study will be linked to an epidemiological survey and molecular analyses of parasite and human genetic polymorphisms. The aims of the study will be to: compare safety, tolerability, and efficacy of combination antimalarial therapies using a longitudinal design; follow plasmodial genetic polymorphisms as longitudinal markers of antimalarial drug resistance; and evaluate the roles of host genetic polymorphisms in antimalarial drug resistance and the incidence of clinical malaria. The clinical study will recruit participants from a defined and mapped source population in the Mulago III Parish, Kawempe District in Kampala, Uganda; conduct a survey of epidemiological factors on participants; and follow clinical care and outcomes over an extended period of time. Molecular analyses of parasite and human genetic polymorphisms will evaluate the impact of parasite mutations on treatment efficacy, the effects of repeated treatments on selection for resistance-mediating genotypes, and the impact of host polymorphisms on the incidence of malaria and responses to therapy. Phase I will include a random sample of 600 Ugandan children between the ages of 1-10 years. Participants will be followed for 3 years for all routine medical care in the study clinic at Mulago Hospital. Children presenting to the study clinic with a new episode of fever will undergo standard evaluation (history, physical examination and Giemsa-stained blood smear) for the diagnosis of malaria. Participants will be randomized to one of three combination treatment regimens at the time of their first diagnosis of uncomplicated malaria. Subsequent episodes of uncomplicated malaria will be treated with each participant's assigned treatment regimen. Clinical treatment failures occurring within 14 days of diagnosis and all episodes of complicated malaria will be treated with quinine, the standard therapy for malaria after treatment failure in Uganda. Routine home visits will be made for participants not seen in the clinic after any consecutive 30-day period. Routine home visits, made every 90 days, will include review of study protocol with the participants, assessment for any outside medical care, a focused history and physical examination and routine laboratory testing. Phase II will be a randomized, open-label, longitudinal clinical trial, comparing two combination antimalarial regimens. Following the first year of follow up, recruitment will be re-opened for children belonging to the same households previously recruited to the study, for children not previously enrolled ages 1-10 years. At this time, all participants will receive an insecticide treated bed net and phase II follow up will begin. All other aspects of subject evaluation, management, and follow-up will be the same as in Phase I, except that researchers will discontinue 30 day finger sticks (subjects will still be visited if they have not been seen in the clinic for 30 days, but finger sticks for blood smears and filter paper will only be performed during clinic evaluations, when clinically indicated or if the patient has not been evaluated in the clinic over a 90 day period). The primary outcome and endpoint (power calculations are based only on this endpoint) for this study will be treatment incidence density (treatments per time at risk) for each treatment arm. Secondary outcomes include drug efficacy and safety and tolerability. Protocol 05-0110 is a sub study of this protocol.

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Age 1 to 10 years.
* Agreement to come to the study clinic for any febrile episode or other illness.
* Agreement to avoid medications administered outside the study.
* Willingness of parents or guardians to provide informed consent.

Phase II

* Child and Guardian/Parent belong to household currently enrolled in the study.
* Age 1 to 10 years.
* Agreement to come to the study clinic for any febrile episode or other illness.
* Agreement to avoid medications administered outside the study.
* Willingness of parents or guardians to provide informed consent.

Exclusion Criteria:

Phase I

* History (obtained from the parent/guardian) of any known serious chronic disease requiring frequent medical care (e.g. AIDS, sickle cell disease, malignancy).
* Intention to move from Kampala during the follow-up period.
* History (obtained from the parent/guardian) of serious side effects to study medications or sulfa drugs.
* Weight < 10 kg
* Severe malnutrition defined as weight-for-height or height-for-age Z-score <-3.
* Homozygous hemoglobin SS (sickle cell) result by hemoglobin electrophoresis.
* Life-threatening screening laboratory value in the absence of malaria:
* Absolute neutrophil count: < 250/mm^3
* Hemoglobin: < 5.0 g/dL
* Platelet count: < 25,000/mm^3
* Creatinine: < 2 years: > 1.5 mg/dL, greater than or equal to 2 years: > 2.0 mg/dL
* ALT: > 15.0 x ULN
* Bilirubin: > 7.5 x ULN Phase II
* History of any known serious chronic disease requiring frequent medical attention (e.g. AIDS, sickle cell disease, malignancy)
* Intention to move from Kampala during the follow-up period
* Any history of serious side effects to study medications
* Weight < 10 kg
* Severe malnutrition
* Life-threatening screening laboratory test result

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 601 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Annual incidence of malaria per treatment arm | duration of study

SECONDARY OUTCOMES:
Short term: clinical and parasitological outcome; rates of fever and parasite clearance; presence of gametocytes following treatment | 14 days
Short term: change in hemoglobin level from day 0-14; safety and tolerability of study medications | 14 days
Long term: risk of reinfection using Kaplan-Meier product limit estimates of risk at various time intervals | Beyond 14 days to end of study
Long term: risk of recrudescence; change in hemoglobin level; safety and tolerability of study medications | Beyond 14 days to end of study
Longitudinal: prevalence of asymptomatic parasitemia; mean hemoglobin | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assessment Center - Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Result] Davis JC, Clark TD, Kemble SK, Talemwa N, Njama-Meya D, Staedke SG, Dorsey G. Longitudinal study of urban malaria in a cohort of Ugandan children: description of study site, census and recruitment. Malar J. 2006 Mar 21;5:18. doi: 10.1186/1475-2875-5-18. PMID 16551365
- [Result] Njama-Meya D, Clark TD, Nzarubara B, Staedke S, Kamya MR, Dorsey G. Treatment of malaria restricted to laboratory-confirmed cases: a prospective cohort study in Ugandan children. Malar J. 2007 Jan 21;6:7. doi: 10.1186/1475-2875-6-7. PMID 17239256
- [Result] Dorsey G, Staedke S, Clark TD, Njama-Meya D, Nzarubara B, Maiteki-Sebuguzi C, Dokomajilar C, Kamya MR, Rosenthal PJ. Combination therapy for uncomplicated falciparum malaria in Ugandan children: a randomized trial. JAMA. 2007 May 23;297(20):2210-9. doi: 10.1001/jama.297.20.2210. PMID 17519410
- [Result] Clark TD, Greenhouse B, Njama-Meya D, Nzarubara B, Maiteki-Sebuguzi C, Staedke SG, Seto E, Kamya MR, Rosenthal PJ, Dorsey G. Factors determining the heterogeneity of malaria incidence in children in Kampala, Uganda. J Infect Dis. 2008 Aug 1;198(3):393-400. doi: 10.1086/589778. PMID 18522503
- [Result] Maiteki-Sebuguzi C, Jagannathan P, Yau VM, Clark TD, Njama-Meya D, Nzarubara B, Talisuna AO, Kamya MR, Rosenthal PJ, Dorsey G, Staedke SG. Safety and tolerability of combination antimalarial therapies for uncomplicated falciparum malaria in Ugandan children. Malar J. 2008 Jun 11;7:106. doi: 10.1186/1475-2875-7-106. PMID 18547415
- [Result] Staedke SG, Jagannathan P, Yeka A, Bukirwa H, Banek K, Maiteki-Sebuguzi C, Clark TD, Nzarubara B, Njama-Meya D, Mpimbaza A, Rosenthal PJ, Kamya MR, Wabwire-Mangen F, Dorsey G, Talisuna AO. Monitoring antimalarial safety and tolerability in clinical trials: a case study from Uganda. Malar J. 2008 Jun 11;7:107. doi: 10.1186/1475-2875-7-107. PMID 18547416
- [Result] Greenhouse B, Slater M, Njama-Meya D, Nzarubara B, Maiteki-Sebuguzi C, Clark TD, Staedke SG, Kamya MR, Hubbard A, Rosenthal PJ, Dorsey G. Decreasing efficacy of antimalarial combination therapy in Uganda is explained by decreasing host immunity rather than increasing drug resistance. J Infect Dis. 2009 Mar 1;199(5):758-65. doi: 10.1086/596741. PMID 19199542
- [Result] Clark TD, Njama-Meya D, Nzarubara B, Maiteki-Sebuguzi C, Greenhouse B, Staedke SG, Kamya MR, Dorsey G, Rosenthal PJ. Incidence of malaria and efficacy of combination antimalarial therapies over 4 years in an urban cohort of Ugandan children. PLoS One. 2010 Jul 30;5(7):e11759. doi: 10.1371/journal.pone.0011759. PMID 20689585